CLINICAL TRIAL: NCT02229539
Title: A Phase III Placebo-Controlled, Randomized Three-Arm Study of Doxepin and a Topical Rinse in the Treatment of Acute Oral Mucositis Pain in Patients Receiving Radiotherapy With or Without Chemotherapy
Brief Title: Doxepin and a Topical Rinse in the Treatment of Acute Oral Mucositis Pain in Patients Receiving Radiotherapy With or Without Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A221304; U10CA037447 (NIH); UG1CA189823 (NIH); NCI-2014-01877 (Registry Identifier: NCI Clinical Trials Reporting Office)
Record Dates: First submitted 2014-08-29; First posted 2014-09-01 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Acute Oral Mucositis Pain
MeSH Terms: interventions — Doxepin; Diphenhydramine; Lidocaine; Antacids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- doxepin rinse (Experimental): Patients receive 2.5 mL (25 mg) doxepin and 2.5 mL water orally. Doxepin rinse is administered in the clinic on Day 1 (Cycle 1). There is an optional continuation phase within seven days following Day 1 (Cycle 1), patients will be encouraged to continue treatment with the study agent for an additional week (Cycle 2) where the patient takes the rinse at home every 4 hours. Chemotherapy is allowed during the continuation phase. Patients randomized to doxepin or placebo, they and their caregivers will continue to be blinded to the treatment.
  Patients will complete the Oral Symptoms booklet per the protocol.
  Interventions: Drug: doxepin hydrochloride oral solution
- DLA (diphenhydramine, lidocaine and antacid) rinse (Active Comparator): Patients receive 5.0 mL DLA orally. DLA is administered in the clinic on Day 1 (Cycle 1). There is an optional continuation phase within seven days following Day 1 (Cycle 1), patients will be encouraged to continue treatment with the study agent for an additional week (Cycle 2) where the patient takes the rinse at home every 4 hours. Chemotherapy is allowed during the continuation phase. Patients receiving DLA during the continuation phase of the study, they and/or caregivers may be aware that they are receiving DLA.
  Patients will complete the Oral Symptoms booklet per the protocol.
  Interventions: Drug: DLA (diphenhydramine, lidocaine and antacids) rinse
- placebo rinse (Placebo Comparator): Patients receive 2.5 mL placebo and 2.5 mL water orally. The placebo rinse is administered in the clinic on Day 1 (Cycle 1). There is an optional continuation phase within seven days following Day 1 (Cycle 1), patients will be encouraged to continue treatment with the study agent for an additional week (Cycle 2) where the patient takes the rinse at home every 4 hours. Chemotherapy is allowed during the continuation phase. Patients randomized to doxepin or placebo, they and their caregivers will continue to be blinded to the treatment.
  Patients will complete the Oral Symptoms booklet per the protocol.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: doxepin hydrochloride oral solution — 2.5 mL (25 mg) doxepin and 2.5 mL water administered orally
  Arms: doxepin rinse
Drug: DLA (diphenhydramine, lidocaine and antacids) rinse — 5.0 mL administered orally
  Arms: DLA (diphenhydramine, lidocaine and antacid) rinse
Other: Placebo — 2.5 mL placebo and 2.5 mL water administered orally
  Arms: placebo rinse

SUMMARY:
The purpose of this study is to test whether a mouthwash made with a drug called doxepin can reduce the pain caused by mouth sores resulting from radiation therapy. A number of mouth rinse preparations exist for patients with treatment-related oral mucositis pain such as the DLA rinse, an over-the-counter medication. This study will evaluate the effects of doxepin compared to DLA (diphenhydramine, lidocaine and antacids) and placebo.Doxepin is approved by the Food and Drug Administration (FDA) for the treatment of depression, anxiety, long-term pain management, as well as management of rash.

DETAILED DESCRIPTION:
Patients are stratified according to sex (male vs. female), concurrent use of chemotherapy (no vs. yes), patient age at registration (< 60 years old vs. ≥ 60 years old and RTOG acute radiation morbidity criteria (1 vs. 2 vs 3 or more). Protocol therapy will consist of 2 cycles. Patients are randomized to one of three treatment regimens, which include doxepin, DLA and placebo. Cycle One will consist of one day. The care provider or nurse will confirm that the oral pain is at least 4 out of 10 severity level at the time of the rinse on the first day of the study. Patient will be asked to complete the baseline evaluation in the Oral Symptoms booklet. If the pain score is less than 4 then administration will be delayed until the pain is at least 4. Cycle Two will consist of an optional continuation phase lasting up to 7 days. Initiation of the Cycle 2/Continuation Phase may be delayed up to one week after Cycle 1/Day 1.

Primary Objective:

1. Determine whether the doxepin rinse or DLA rinse is more effective than placebo in reducing OM-related pain in patients undergoing RT to the oral cavity, as measured by a patient-reported questionnaire at baseline, 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, and 4 hours.

Secondary Objectives:

1. Assess the adverse event profile of the doxepin rinse, the DLA rinse agent, and the placebo using a patient-reported questionnaire at 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, and 4 hours for domains of unpleasant taste, burning or stinging discomfort, and drowsiness.
2. Compare the incidence of using additional analgesics between 1 and 4 hours after the initial mouthwash, between the doxepin oral rinse, the DLA rinse agent, and the placebo arms.
3. Compare the length of time that each study product is used by patients in the one-week continuation phase.
4. Compare the daily pain scores in the one-week continuation phase for the three study arms.
5. Compare the 24-hour morphine equivalent dose used in the continuation phase for the three study arms.

ELIGIBILITY:
1. Documentation of Disease: Histologic documentation of malignancy currently undergoing a course of RT (with or without chemotherapy) including the oral cavity and/or oropharyngeal area to a dose of at least 4500 cGy using more than 5 fractions (i.e., stereotactic body radiation therapy [SBRT] is not allowed).
2. Physical exam demonstrating evidence of radiotherapy-related mucositis in the visible oral cavity and/or oropharynx consistent with mucous membrane toxicity greater than 0 using the Acute Radiation Morbidity Scoring Criteria.
3. At least 4 (out of 10) patient-reported oral pain related to oral mucositis secondary to RT for which the patient seeks relief, as measured on the Oral Pain Assessment.

   Note: The pain score must be at least 4 at the time that the patient starts the first dose of study medication. The patient may be enrolled to the study if s/he, at times, has a pain score of at least 4, so long as initiation of study treatment begins when the pain score is at least 4.
4. Ability to complete questionnaire(s) by themselves or with assistance.
5. No known allergy to diphenhydramine, lidocaine, antacid (aluminum hydroxide, magnesium hydroxide, and simethicone), doxepin, tricyclic antidepressants, or any known component of the drug formulation in the testing arms.
6. No use of any anti-arrhythmic medication (except for beta-blockers) including lidocaine, linezolid, ipratropium, or medications with high anti-cholinergic potency (including neostigmine, a tricyclic antidepressant or a monoamine oxidase inhibitor) within 2 weeks prior to registration.
7. No current diagnosed untreated or unresolved oral candidiasis or oral HSV infection.
8. No history of untreated narrow angle glaucoma within 6 weeks prior to registration.
9. No untreated urinary retention within 6 weeks prior to registration.
10. No current use of glutamine or sucralfate powders at the time of registration (no washout required).
11. No cryotherapy for prophylactic mucosal protection within 6 weeks prior to registration.
12. Not pregnant, because patients eligible for this study will be receiving radiotherapy, which has known genotoxic, mutagenic and teratogenic effects. Therefore, for women of childbearing potential only, a negative pregnancy test done ≤ 28 days prior to registration is required.
13. Age ≥ 18 years
14. ECOG Performance Status 0, 1, or 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2016-05-23 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Miller, MD, MS, Study Chair — Mayo Clinic
Locations (349):
- United States (349):
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute CCOP, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare- Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center Radiation Oncology Service at the Central Illinois Comprehensive CC, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas - Independence, Independence, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas - Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Maine Medical Center - Bramhall Campus, Portland, Maine
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Central Care Center - Carrie J. Babb Cancer Center, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Cox Health South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute - South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Henderson, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Cancer and Blood Specialists-Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Veterans Affairs Western New York Health Care System-Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore-LIJ Health System/Center for Advanced Medicine, New Hyde Park, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Carolina Surgical Clinic of Charlotte PA, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Lake Norman Hematology Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Novant Health Oncology Specialists-Kernersville, Kernersville, North Carolina
  - Novant Health Oncology Specialists-Davidson County, Lexington, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Lake Norman Hematology Oncology Specialists-Mooresville, Mooresville, North Carolina
  - Novant Health Oncology Specialists-Mount Airy, Mount Airy, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Carolina Oncology Associates PA, Salisbury, North Carolina
  - Novant Health Oncology Specialists-Statesville, Statesville, North Carolina
  - Novant Health Oncology Specialists-Wilkesboro, Wilkesboro, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Winston-Salem Health Care, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazelton, Hazleton, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Greenville Health System Cancer Institute - Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Avera Saint Luke's Hospital and Cancer Center, Aberdeen, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Medical Center - Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint John Medical Center, Longview, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Westfields Hospital/Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Door County Cancer Center, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Saint Clare's Hospital, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming

REFERENCES:
- [Derived] Sio TT, Le-Rademacher JG, Leenstra JL, Loprinzi CL, Rine G, Curtis A, Singh AK, Martenson JA Jr, Novotny PJ, Tan AD, Qin R, Ko SJ, Reiter PL, Miller RC. Effect of Doxepin Mouthwash or Diphenhydramine-Lidocaine-Antacid Mouthwash vs Placebo on Radiotherapy-Related Oral Mucositis Pain: The Alliance A221304 Randomized Clinical Trial. JAMA. 2019 Apr 16;321(15):1481-1490. doi: 10.1001/jama.2019.3504. PMID 30990550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two-hundred and seventy-five participants (92 Doxepin, 91 DLA and 92 Placebo) were enrolled between November 2014 to May 2016. Data as of 8/21/2017 was summarized and reported.
Pre-assignment Details: Total of 45 participants were excluded from all analyses due to 23 cancellations, 19 with mouth pain score<4 prior to treatment, 1 ineligible, 1 did not return questionnaire booklet and 1 inadvertently unblinding by study team.
Groups:
- Doxepin: Patients receive 2.5 mL (25 mg) doxepin and 2.5 mL water orally in the clinic on Day 1 (Cycle 1). Patients will be encouraged to continue treatment with the study agent for an additional week (Cycle 2).
- DLA (Diphenhydramine, Lidocaine and Antacid): Patients receive 5.0 mL DLA orally in the clinic on Day 1 (Cycle 1). Patients will be encouraged to continue treatment with the study agent for an additional week (Cycle 2).
- Placebo: Patients receive 2.5 mL placebo and 2.5 mL water orally in the clinic on Day 1 (Cycle 1). Patients will be encouraged to continue treatment with the study agent for an additional week (Cycle 2).
Period: Cycle 1 (Treatment Per Protocol)
Arm/Group | Doxepin | DLA (Diphenhydramine, Lidocaine and Antacid) | Placebo
Started | 78 | 76 | 76
Completed | 78 | 75 | 74
Not Completed | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Alternate Therapy | 0 | 0 | 1
Not completed — Medical Problems | 0 | 0 | 1
Period: Cycle 2 (Optional Continuation Phase)
Arm/Group | Doxepin | DLA (Diphenhydramine, Lidocaine and Antacid) | Placebo
Started (Include only those who completed cycle 1 and chose to continue the study drug for up to 7 days.) | 35 | 38 | 32
Completed | 28 | 31 | 22
Not Completed | 7 | 7 | 10
Not completed — Withdrawal by Subject | 5 | 6 | 8
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Alternative Therapy | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All participants who met eligibility criteria, had mouth pain score of at least 4 on 0 to 10 scale with higher scores indicated worst pain and started the treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxepin | DLA (Diphenhydramine, Lidocaine and Antacid) | Placebo | Total
Number analyzed (Participants) | 78 | 76 | 76 | 230
Age, Continuous [Median (Full Range); unit: years] | 61.5 [26 to 87] | 60.0 [23 to 82] | 60.0 [31 to 94] | 60 [23 to 94]
Age, Customized [Count of Participants; unit: Participants]
  <60 years old | 35 | 34 | 37 | 106
  >=60 years old | 43 | 42 | 39 | 124
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 19 | 56
  Male | 59 | 58 | 57 | 174
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 7 | 4 | 13
  White | 75 | 67 | 71 | 213
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 78 | 76 | 76 | 230
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0=Asymptomatic and fully active | 37 | 31 | 33 | 101
  1=Symptomatic and fully ambulatory | 40 | 39 | 40 | 119
  2=Symptomatic, <50% in bed during the day | 1 | 6 | 3 | 10
Concurrent use of chemotherapy [Count of Participants; unit: Participants]
  Yes | 62 | 62 | 64 | 188
  No | 16 | 14 | 12 | 42
Mucous Membrane Grade [Count of Participants; unit: Participants] — Mucous membrane grade:>
  >> 0=no change over baseline, 1=injection/may experience mild pain not requiring analgesic, 2=patchy mucositis which may produce an inflammatory serosanguinitis discharge/ may experience moderate pain requiring analgesia, 3=confluent fibrinous mucositis/ may include severe pain requiring narcotic, 4=Ulceration, hemorrhage or necrosis.
  Participants
    1 | 17 | 16 | 16 | 49
    2 | 47 | 48 | 49 | 144
    3 or more | 14 | 12 | 11 | 37

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Curve (AUC) of Total Pain Reduction
Description: Total pain reduction (mouth and throat) was measured by the numerical analogue scale of mouth pain on a scale of 0 to 10, with 0=no pain and 10=worst pain in the questionnaires taken at baseline, and 5, 15, 30, 60, 120, 240 minutes after assigned treatment for doxepin or DLA vs. placebo. The total pain reduction was calculated by the (average of mouth and throat) area under the curve (AUC) adjusting for baseline, with time scale (baseline, 5, 15, 30, 60, 120 and 240 minutes post treatment) replaced by a numerical scale of 0, 1, 2, 3, 4, 5 and 6 respectively. The AUC was prorated when there are terminal missing data. If the missing data were intermittent, simple imputation by trapezoidal rules were applied to calculate the AUC. If a patient cancelled, was missing baseline data, or only provided baseline data, he/she was excluded from the statistical analysis.
Time Frame: Baseline, 5, 15, 30, 60, 120, 240 minutes post treatment
Population: All participants who met eligibility criteria, had mouth pain score of at least 4 on 0 to 10 scale with higher scores indicated worst pain and started the treatment and had mouth and throat pain data at baseline and at least one time point beyond baseline.
Measure: Mean (Standard Deviation); unit: units on a scale*time scale
Arm/Group | Doxepin | DLA (Diphenhydramine, Lidocaine and Antacid) | Placebo
Number analyzed (Participants) | 78 | 76 | 76
units on a scale*time scale | 11.6 (9.7) | 11.7 (8.1) | 8.7 (9.9)
Statistical Analysis 1: Comparison: Doxepin vs Placebo; Test type: Superiority or Other; p = 0.02, Wilcoxon rank-sum
Statistical Analysis 2: Comparison: DLA (Diphenhydramine, Lidocaine and Antacid) vs Placebo; Test type: Superiority or Other; p = 0.004, Wilcoxon rank-sum

2. Secondary Outcome: Area Under the Curve (AUC) of Total Unpleasant Taste of the Oral Rinse
Description: Total unpleasant taste was measured by the numerical analogue scale of taste of the oral rinse on a scale of 0 to 10, with 0=acceptable and 10=terrible in the questionnaires taken at 5, 15, 30, 60, 120, 240 minutes after assigned treatment for doxepin or DLA vs. placebo. The total unpleasant taste was calculated by the area under the curve (AUC) adjusting for 5 minutes post treatment, with time scale (5, 15, 30, 60, 120 and 240 minutes post treatment) replaced by a numerical scale of 1, 2, 3, 4 5 and 6 respectively. The AUC was prorated when there are terminal missing data. If the missing data were intermittent, simple imputation by trapezoidal rules were applied to calculate the AUC. If a patient cancelled, was missing 5 minutes after treatment data, or only provided 5 minutes after treatment data, he/she was excluded from the statistical analysis.
Time Frame: 5, 15, 30, 60, 120, 240 minutes post treatment
Measure: Median (Inter-Quartile Range); unit: units on a scale*units on a scale
Arm/Group | Doxepin | DLA (Diphenhydramine, Lidocaine and Antacid) | Placebo
Number analyzed (Participants) | 78 | 76 | 76
units on a scale*units on a scale | 3.5 [0 to 8.5] | 2.0 [0 to 6.3] | 0.8 [0 to 3.0]

3. Secondary Outcome: Area Under the Curve (AUC) of Total Stinging or Burning From the Oral Rinse
Description: Total stinging or burning was measured by the numerical analogue scale of stinging or burning from the oral rinse on a scale of 0 to 10, with 0=no stinging or burning and 10=worst stinging or burning possible in the questionnaires taken at 5, 15, 30, 60, 120, 240 minutes after assigned treatment for doxepin or DLA vs. placebo. The total stinging or burning was calculated by the area under the curve (AUC) adjusting for 5 minutes post treatment, with time scale (5, 15, 30, 60, 120 and 240 minutes post treatment) replaced by a numerical scale of 1, 2, 3, 4 5 and 6 respectively. The AUC was prorated when there are terminal missing data. If the missing data were intermittent, simple imputation by trapezoidal rules were applied to calculate the AUC. If a patient cancelled, was missing 5 minutes after treatment data, or only provided 5 minutes after treatment data, he/she was excluded from the statistical analysis.
Time Frame: 5, 15, 30, 60, 120, 240 minutes post treatment
Measure: Median (Inter-Quartile Range); unit: units on a scale*units on a scale
Arm/Group | Doxepin | DLA (Diphenhydramine, Lidocaine and Antacid) | Placebo
Number analyzed (Participants) | 78 | 76 | 76
units on a scale*units on a scale | 5.3 [2.5 to 11.0] | 0.8 [0 to 4.8] | 0.5 [0 to 3.0]

4. Secondary Outcome: Area Under the Curve (AUC) of Total Drowsiness
Description: Total drowsiness was measured by the numerical analogue scale of drowsiness on a scale of 0 to 10, with 0=no drowsiness and 10=extreme drowsiness, leading to sleep in the questionnaires taken at baseline, and 5, 15, 30, 60, 120, 240 minutes after assigned treatment for doxepin or DLA vs. placebo. The total drowsiness was calculated by the area under the curve (AUC) adjusting for baseline, with time scale (baseline, 5, 15, 30, 60, 120 and 240 minutes post treatment) replaced by a numerical scale of 0, 1, 2, 3, 4, 5 and 6 respectively. The AUC was prorated when there are terminal missing data. If the missing data were intermittent, simple imputation by trapezoidal rules were applied to calculate the AUC. If a patient cancelled, was missing baseline data, or only provided baseline data, he/she was excluded from the statistical analysis.
Time Frame: Baseline, 5, 15, 30, 60, 120, 240 minutes post treatment
Measure: Median (Inter-Quartile Range); unit: units on a scale*units on a scale
Arm/Group | Doxepin | DLA (Diphenhydramine, Lidocaine and Antacid) | Placebo
Number analyzed (Participants) | 78 | 76 | 76
units on a scale*units on a scale | 0 [-2.5 to 3.0] | -1.8 [-7.3 to 0] | 0 [-8.0 to 0]

5. Secondary Outcome: The Incidence of Using Alternative Analgesics
Description: Patients were asked if they have taken any other pain medications, if yes, to record the name, strength and when they have taken the pain medications in the 120 minutes and 240 minutes post treatment questionnaires.
Time Frame: At 120 and 240 minutes post treatment
Population: Some patients are missing their Additional Analgesic Use. All participants who met eligibility criteria, had mouth pain score of at least 4 on 0 to 10 scale with higher scores indicated worst pain and started the treatment and has responded to the question about if they have taken any other pain medications at the indicated time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Doxepin | DLA (Diphenhydramine, Lidocaine and Antacid) | Placebo
Number analyzed (Participants) | 78 | 76 | 76
Participants
  120 minutes: number analyzed (Participants) | 77 | 73 | 70
  120 minutes | 10 | 7 | 14
  240 minutes: number analyzed (Participants) | 76 | 72 | 72
  240 minutes | 13 | 14 | 21

6. Secondary Outcome: Patient Preference for Continued Therapy With Oral Rinse After Initial Test Rinse Phase
Description: Patients were asked: "Based on your experience with this current oral rinsing medication, would you want to take another dose now if it were available?" in the 240 minutes post treatment questionnaire.
Time Frame: At 240 minutes post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Doxepin | DLA (Diphenhydramine, Lidocaine and Antacid) | Placebo
Number analyzed (Participants) | 75 | 73 | 71
Participants | 45 | 46 | 38

7. Secondary Outcome: Frequency of Study Rinse Used in the Continuation Phase
Description: Patients were asked: "Did you use the study rinse today?" daily questionnaire during the optional continuation phase (Cycle 2).
Time Frame: Up to 7 days.
Population: All participants who met eligibility criteria, had mouth pain score of at least 4 on 0 to 10 scale with higher scores indicated worst pain, completed the cycle 1 treatment, has started treatment in the optional continuation phase and has responded to the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Doxepin | DLA (Diphenhydramine, Lidocaine and Antacid) | Placebo
Number analyzed (Participants) | 35 | 38 | 32
Participants
  Cycle 2 Day 1: number analyzed (Participants) | 35 | 37 | 31
  Cycle 2 Day 1: Yes | 33 | 37 | 30
  Cycle 2 Day 1: No | 2 | 0 | 1
  Cycle 2 Day 2: number analyzed (Participants) | 34 | 36 | 28
  Cycle 2 Day 2: Yes | 30 | 33 | 25
  Cycle 2 Day 2: No | 4 | 3 | 3
  Cycle 2 Day 3: number analyzed (Participants) | 34 | 35 | 27
  Cycle 2 Day 3: Yes | 30 | 27 | 22
  Cycle 2 Day 3: No | 4 | 8 | 5
  Cycle 2 Day 4: number analyzed (Participants) | 32 | 33 | 25
  Cycle 2 Day 4: Yes | 29 | 25 | 18
  Cycle 2 Day 4: No | 3 | 8 | 7
  Cycle 2 Day 5: number analyzed (Participants) | 32 | 30 | 24
  Cycle 2 Day 5: Yes | 27 | 24 | 17
  Cycle 2 Day 5: No | 5 | 6 | 7
  Cycle 2 Day 6: number analyzed (Participants) | 32 | 30 | 21
  Cycle 2 Day 6: Yes | 27 | 26 | 14
  Cycle 2 Day 6: No | 5 | 4 | 7
  Cycle 2 Day 7: number analyzed (Participants) | 30 | 31 | 22
  Cycle 2 Day 7: Yes | 24 | 25 | 15
  Cycle 2 Day 7: No | 6 | 6 | 7

8. Secondary Outcome: Median Mouth Pain Score in the Continuation Phase
Description: Mouth pain scores was measured using the numerical analogue scale ranging from scale of 0 to 10, with 0=no pain and 10=worst pain daily during the optional continuation phase (Cycle 2).
Time Frame: Day 1 to Day 7 in the Continuation Phase
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Doxepin | DLA (Diphenhydramine, Lidocaine and Antacid) | Placebo
Number analyzed (Participants) | 35 | 38 | 32
units on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 34 | 36 | 31
  Cycle 2 Day 1 | 6.0 [0.0 to 9.0] | 5.5 [1.0 to 9.0] | 5.0 [1.0 to 9.0]
  Cycle 2 Day 2: number analyzed (Participants) | 34 | 36 | 26
  Cycle 2 Day 2 | 5.0 [0.0 to 9.0] | 5.5 [1.0 to 8.0] | 5.0 [1.0 to 9.0]
  Cycle 2 Day 3: number analyzed (Participants) | 33 | 35 | 24
  Cycle 2 Day 3 | 5.0 [0.0 to 10.0] | 5.0 [1.0 to 8.0] | 5.0 [1.0 to 9.0]
  Cycle 2 Day 4: number analyzed (Participants) | 30 | 33 | 22
  Cycle 2 Day 4 | 5.0 [0.0 to 9.0] | 5.0 [1.0 to 9.0] | 5.0 [2.0 to 9.0]
  Cycle 2 Day 5: number analyzed (Participants) | 31 | 30 | 22
  Cycle 2 Day 5 | 5.0 [0.0 to 9.0] | 5.0 [1.0 to 8.0] | 5.0 [0.0 to 9.0]
  Cycle 2 Day 6: number analyzed (Participants) | 30 | 31 | 21
  Cycle 2 Day 6 | 5.5 [0.0 to 9.0] | 5.0 [1.0 to 9.0] | 4.0 [2.0 to 9.0]
  Cycle 2 Day 7: number analyzed (Participants) | 25 | 29 | 20
  Cycle 2 Day 7 | 5.0 [0.0 to 9.0] | 5.0 [1.0 to 8.0] | 4.5 [2.0 to 10.0]

9. Secondary Outcome: The Incidence of Using Alternative Analgesics in the Continuation Phase
Description: Patients were asked if they have taken any medications for pain over the past 24 hours, if yes, to record the name, strength and when they have taken the pain medications daily during the optional continuation phase (Cycle 2).
Time Frame: Day 1 to Day 7 in the Continuation Phase
Population: All participants who met eligibility criteria, had mouth pain score of at least 4 on 0 to 10 scale with higher scores indicated worst pain and started the treatment and has responded to the question about if they have taken any other pain medications at the indicated time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Doxepin | DLA (Diphenhydramine, Lidocaine and Antacid) | Placebo
Number analyzed (Participants) | 35 | 38 | 32
Participants
  Cycle 2 Day 1: number analyzed (Participants) | 34 | 35 | 31
  Cycle 2 Day 1: Yes | 22 | 20 | 21
  Cycle 2 Day 1: No | 12 | 15 | 10
  Cycle 2 Day 2: number analyzed (Participants) | 33 | 36 | 27
  Cycle 2 Day 2: Yes | 19 | 22 | 19
  Cycle 2 Day 2: No | 14 | 14 | 8
  Cycle 2 Day 3: number analyzed (Participants) | 33 | 34 | 24
  Cycle 2 Day 3: Yes | 17 | 19 | 17
  Cycle 2 Day 3: No | 16 | 15 | 7
  Cycle 2 Day 4: number analyzed (Participants) | 31 | 32 | 23
  Cycle 2 Day 4: Yes | 20 | 22 | 16
  Cycle 2 Day 4: No | 11 | 10 | 7
  Cycle 2 Day 5: number analyzed (Participants) | 29 | 30 | 22
  Cycle 2 Day 5: Yes | 19 | 16 | 15
  Cycle 2 Day 5: No | 10 | 14 | 7
  Cycle 2 Day 6: number analyzed (Participants) | 30 | 31 | 21
  Cycle 2 Day 6: Yes | 22 | 20 | 14
  Cycle 2 Day 6: No | 8 | 11 | 7
  Cycle 2 Day 7: number analyzed (Participants) | 25 | 30 | 19
  Cycle 2 Day 7: Yes | 17 | 19 | 13
  Cycle 2 Day 7: No | 8 | 11 | 6

ADVERSE EVENTS:
Time Frame: In clinic at 5, 15, 30, and 60 minutes after oral rinse and daily for up to 7 days, beginning within 1 week of Day 1.
Description: All participants who met eligibility criteria, had mouth pain score of at least 4 on 0 to 10 scale with higher scores indicated worst pain, started the treatment and had adverse events assessed during the reporting period. Adverse events were not assessed on six participants (2 DLA and 4 Placebo).
Arm/Group | Doxepin | Placebo | DLA (Diphenhydramine, Lidocaine and Antacid)
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 2/78 | 3/72 | 3/74
Other Adverse Events (participants affected / at risk) | 17/78 | 7/72 | 8/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxepin (N=78) | Placebo (N=72) | DLA (Diphenhydramine, Lidocaine and Antacid) (N=74)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxepin (N=78) | Placebo (N=72) | DLA (Diphenhydramine, Lidocaine and Antacid) (N=74)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 1 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2)
Oral dysesthesia (Gastrointestinal disorders) | 3 (3) | 2 (3) | 3 (3)
Oral pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 6 (7) | 1 (1) | 2 (3)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (3) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 3 (4) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Body odor (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less